CLINICAL TRIAL: NCT02734407
Title: Long-Term Efficacy and Safety of Aflibercept Intravitreal Injections for the Treatment of Diabetic Macular Edema in Subjects Who Completed the Three Year VISTA-DME Trial
Brief Title: Long-Term Efficacy and Safety of Aflibercept Intravitreal Injections for the Treatment of Diabetic Macular Edema
Acronym: Endurance3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Retina-Vitreous Associates Medical Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endurance 3
Record Dates: First submitted 2014-12-16; First posted 2016-04-12 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Clinically Significant Diabetic Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-Label Arm (Experimental): 2mg Aflibercept, as needed, intravitreal administration.
  All subjects will be treated with intravitreal (IVT) aflibercept injections as needed in the presence of clinically relevant diabetic macular edema (CR-DME). If CR-DME is not present the subject will not receive an IVT aflibercept injection and will be observed.
  If a subject has recurrent CR-DME they will receive an IVT aflibercept 2.0 mg injection and interval between visits will be reduced to 4 weeks.
  At week 12 through end of study, all subjects will be evaluated for focal laser treatment.
  Interventions: Procedure: Assigned Intervention; Drug: aflibercept 2.0 mg

INTERVENTIONS:
Procedure: Assigned Intervention — All subjects receiving PRN IVT aflibercept injections will be evaluated for focal laser treatment beginning at week 12 through the end of the study as assigned intervention. If the subject meets any of the criteria for focal laser treatment (FLT), fluorescein angiography (FA) will be performed to guide the focal laser treatment. Focal laser treatment and focal laser re-treatment will be administered no more than once every 90 days.
  Other Names: FLT
Drug: aflibercept 2.0 mg — If a subject has recurrent CR-DME they will receive an IVT aflibercept injection
  Other Names: Eylea; VEGF-Trap

SUMMARY:
The Endurance Trial is a Phase IV open label clinical study to assess the need for ongoing intravitreal aflibercept injections after the 3-year VISTA DME (VGFT-OD-1009) endpoint. Subjects will be treated with intravitreal aflibercept injections pro re nata (PRN) based on the presence of CR-DME (Clinically Relevant-DME). In addition, subjects who meet re-treatment criteria will be eligible for focal laser treatment every 90 days

DETAILED DESCRIPTION:
The Endurance3 Trial is a Phase IV open label study to assess the need for ongoing intravitreal aflibercept injections after the 3 year VISTA DME (VGFT-OD-1009) endpoint. Subjects will be treated with intravitreal aflibercept injections pro re nata (PRN) upon the presence of CR-DME (Clinically Relevant DME) as noted by OCT (Optical Coherence Tomography) imaging and examination. In addition, subjects who meet the re-treatment criteria will be eligible for focal laser treatment every 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled and completed VISTA DME (VGFT-OD-1009) clinical trial
* Willing and able to comply with clinic visits and study-related procedures
* Provide signed informed consent
* Enrollment in the trial within 12 weeks of trial activation

Exclusion Criteria:

* Prior treatment with anti-VEGF therapy in the study eye within 28 days of baseline
* Pregnant or breast-feeding women
* Sexually active ment or women of childbearing potential who are unwilling to practice adequate contraception during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-01; Primary Completion 2017-09-27 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
Mean number of intravitreal aflibercept injections in 52 weeks | 12 months
Proportion of subjects receiving 0 aflibercept injections in 52 weeks | 12 months
Longer-term efficacy of aflibercept intravitreal injections as assessed by the mean number of injections in 52 weeks | 12 months
Safety of ongoing aflibercept intravitreal injections as assessed by the incidence and severity of ocular and systemic adverse events | 12 months

SECONDARY OUTCOMES:
Vision Change | 12 months
  Mean change in visual acuity from baseline to week 52
Vision loss | 12 months
  Proportion of subjects with gain or loss of 0 to 5 letters from baseline to week 52
Change in central retinal thickness | 12 months
  Mean change in central retinal thickness from baseline to week 52
Development of clinically relevant diabetic macular edema | 12 months
  Percentage of subjects with no clinically relevant diabetic macular edema seen on SD-OCT from baseline to week 52
Evaluation of Diabetic Retinopathy (Proportion of subjects with stable, worsened, or improved diabetic retinopathy as identified by eye examination and imaging) | 12 months
  Proportion of subjects with stable, worsened, or improved diabetic retinopathy as identified by eye examination and imaging
Role of focal laser treatment in management of DME (Proportion of subjects that receive focal laser treatment and mean number of intravitreal aflibercept injections before and after receiving focal laser treatment) | 12 months
  Proportion of subjects that receive focal laser treatment and mean number of intravitreal aflibercept injections before and after receiving focal laser treatment
Ocular and systemic adverse events | 12 months
  Incidence and severity of ocular and systemic adverse events as identified by eye examinations, imaging, and subject reporting

CONTACTS AND LOCATIONS:
Overall Officials: David Boyer, MD, Principal Investigator — Retina-Vitreous Associates Medical Group